CLINICAL TRIAL: NCT01626209
Title: A Phase I Study of BKM120, Administered Orally in Adult Chinese Patients With Advanced Solid Tumors
Brief Title: A Phase I Study of BKM120 in Adult Chinese Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBKM120Z2102
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2015-02

CONDITIONS: Advanced Breast Cancer, Advanced Carcinomas With Squamous Cell Histology
Keywords: Breast cancer, NSCLC, SCCHN, esophageal cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms | interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BKM120 at: 80 and 100mg/day dose levels (Experimental)
  Interventions: Drug: BKM120

INTERVENTIONS:
Drug: BKM120 — This is a single arm study, with a starting dose of BKM120 at 80mg/day. Two dose levels: 80mg/day and 100mg /day will be tested in the dose escalation phase. At least 3 patients will be enrolled at each dose level and at least 6 evaluable patients required to be treated at the recommended Phase II dose(RP2D)/MTD dose. After dose escalation the 80mg/day and the 100mg /day dose levels will be expanded to evaluate up to approximately a total of 15 patients each (if 100mg is determined as the RP2D/MTD).

SUMMARY:
Dose escalation study with a dose expansion phase, to evaluate safety, tolerability, pharmacokinetics and preliminary efficacy of two dose levels of BKM120 when administered orally.

DETAILED DESCRIPTION:
This is a single arm study, with a starting dose of BKM120 at 80mg/day. Two dose levels: 80mg/day and 100mg /day will be tested in the dose escalation phase. At least 3 patients will be enrolled at each dose level and at least 6 evaluable patients required to be treated at the recommended Phase II dose(RP2D)/MTD dose. After dose escalation the 80mg/day and the 100mg /day dose levels will be expanded to evaluate up to approximately a total of 15 patients each (if 100mg is determined as the RP2D/MTD).

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically-confirmed, advanced unresectable breast cancer or advanced carcinoma with squamous cell histology (including NSCLC, SCCHN, and esophageal) who have progressed on (or not been able to tolerate) standard therapy or for whom no standard anticancer therapy exists
* Patient must provide a representative archival or fresh tumor biopsy for shipping to a Novartis designated laboratory for profiling. Note: one block or ≥ 15 unstained slides is required to determine the PI3K activation status. Whenever possible ≥ 20 unstained slides is preferred.
* Patient has measurable and/or non-measurable disease as per RECIST v1.1 guidelines for solid tumors
* Patient is an adult (female or male) ≥ 18 years of age on the day of consent signature
* Patient has an Eastern Cooperative Oncology Group performance status (ECOG PS) ≤ 2

Exclusion Criteria:

* Patient has received previous treatment with a PI3K inhibitor
* Patient has symptomatic CNS metastases
* Patients with asymptomatic CNS metastases may participate in this trial. The patient must have completed any prior local treatment for CNS metastases ≥ 14 days prior to the start of study treatment (including radiotherapy and/or surgery). If the patient is receiving ongoing corticosteroid therapy, the following criteria must be met:
* The patient must be receiving a stable or decreasing dose ≤ dexamethasone 4 mg/day or equivalent anti-inflammatory potency of another corticosteroid
* The dose of corticosteroid may not have been escalated for at least 14 days before the start of study treatment
* Patient is currently receiving increasing or chronic treatment with corticosteroids (>dexamethasone 4 mg or equivalent anti-inflammatory potency of another corticosteroid) or another immunosuppressive agent.
* Note: Topical applications (e.g., rash), inhaled sprays (e.g., obstructive airways diseases), eye drops or local injections (e.g., intra-articular) are allowed. Patients with previously treated and asymptomatic brain metastases, are permitted to use corticosteroids as per specific protocol criteria
* Patient is currently receiving treatment with drugs known to be moderate or strong inhibitors or inducers of isoenzyme CYP3A. The patient must have discontinued strong inducers for at least one week and must have discontinued strong inhibitors before the treatment is initiated. Switching to a different medication prior to starting study treatment is allowed.

  * Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | During Cycle 1 (28 days)
  An adaptive Bayesian logistic regression model (BLRM) for dose escalation with overdose control will guide the dose escalation. The recommended dose is the one with the highest posterior probablity of DLT in the target interval(16%,33%) among the doses fulfilling the overdose criterion that there is less than 25 % chance of excessive toxicity. A clinical synthesis of the available toxicity information including adverse event that are not DLTs, Pharmacokinetics, Pharmacodynamics, efficacy as well as the recommnendations from the BLRM will be used to determine the dose.

SECONDARY OUTCOMES:
Type, frequency and severity of of Adverse Events (AEs) (based on CTCAE version 4.03 | On a continous basis up to when patient discontinues for progression or until any discontinuation criteria are met e.g AE, patient withdraws consent, Investigator decision; up to 30 days post last study dose
Laboratory and vital sign parameters | Every week cycle 1 & 2 then monthly up to when patient discontinues for progression or until any discontinuation criteria are met e.g AE, patient withdraws consent, Investigator decision,
Pharmacokinetics: plasma concentration-time profiles of BKM120 for Cmax | Day 1 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) Day 8 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) and Day 28 (predose, postdose: 0.5,1,1.5,2,3,4,6,8,24 hr)
Pharmacokinetics: plasma concentration-time profiles of BKM120 for Tmax | Day 1 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) Day 8 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) and Day 28 (predose, postdose: 0.5,1,1.5,2,3,4,6,8,24 hr)
Pharmacokinetics: plasma concentration-time profiles of BKM120 for AUCtlast | Day 1 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) Day 8 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) and Day 28 (predose, postdose: 0.5,1,1.5,2,3,4,6,8,24 hr)
Pharmacokinetics: plasma concentration-time profiles of BKM120 for AUCtau | Day 1 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) Day 8 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) and Day 28 (predose, postdose: 0.5,1,1.5,2,3,4,6,8,24 hr)
Pharmacokinetics: plasma concentration-time profiles of BKM120 for AUCinf | Day 1 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) Day 8 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) and Day 28 (predose, postdose: 0.5,1,1.5,2,3,4,6,8,24 hr)
Pharmacokinetics: plasma concentration-time profiles of BKM120 for AUC%Extrap | Day 1 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) Day 8 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) and Day 28 (predose, postdose: 0.5,1,1.5,2,3,4,6,8,24 hr)
Pharmacokinetics: plasma concentration-time profiles of BKM120 for CL/F | Day 1 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) Day 8 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) and Day 28 (predose, postdose: 0.5,1,1.5,2,3,4,6,8,24 hr)
Pharmacokinetics: plasma concentration-time profiles of BKM120 for Racc | Day 1 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) Day 8 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) and Day 28 (predose, postdose: 0.5,1,1.5,2,3,4,6,8,24 hr)
Pharmacokinetics: plasma concentration-time profiles of BKM120 for T1/2acc | Day 1 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) Day 8 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) and Day 28 (predose, postdose: 0.5,1,1.5,2,3,4,6,8,24 hr)
Pharmacokinetics: plasma concentration-time profiles of BKM120 for Vss/F | Day 1 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) Day 8 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) and Day 28 (predose, postdose: 0.5,1,1.5,2,3,4,6,8,24 hr)
Pharmacokinetics: plasma concentration-time profiles of BKM120 for Rsqadj | Day 1 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) Day 8 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) and Day 28 (predose, postdose: 0.5,1,1.5,2,3,4,6,8,24 hr)
Pharmacokinetics: plasma concentration-time profiles of BKM120 for other PK parameters | Day 1 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) Day 8 (predose, postdose : 0.5,1,1.5,2,3,4,6,8,24 hr) and Day 28 (predose, postdose: 0.5,1,1.5,2,3,4,6,8,24 hr)
Objective Response Rate (ORR) | Every 8 weeks up to when patient discontinues for progression or until any other discontinuation criteria are met e.g AE, patient withdraws consent, Investigator decision
  Evaluated with CT/MRI according to RECIST criteria (RECIST guidelines version 1.1)
Time to Progression (TTP) | Every 8 weeks up to when patient discontinues for progression or until any other discontinuation criteria are met e.g AE, patient withdraws consent, Investigator decision
  Evaluated with CT/MRI according to RECIST criteria (RECIST guidelines version 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- China (3):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou

REFERENCES:
- See also: Results for CBKM120Z2102 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13643